CLINICAL TRIAL: NCT05233735
Title: An Enhanced Transcutaneous Delivery of Topical Betamethasone for the Treatment of Vitiligo Disease
Brief Title: Enhanced Transcutaneous Delivery of Betamethasone for the Treatment of Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Eli Sprecher, MD, MD, PhD, MBA, Tel-Aviv Sourasky Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0853-20
Record Dates: First submitted 2021-10-05; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Vitiligo
Keywords: Vitiligo; Tixel; Enhanced Transcutaneous Delivery
MeSH Terms: conditions — Vitiligo | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Recruited patients will have at least 3 × 3 cm patches in greatest dimensions in symmetrical locations for example both forearms, both legs ect. one side will serve as target lesion and the other willl rec. Patients receiving topical or systemic therapy for vitiligo will be kept off treatment for 4 weeks prior to start of therapy.
  each patient will have 2 different treatments. one side - topical application of Betamethasone alone other side - enhanced Transcutaneous Delivery of Topical Betamethasone for the Treatment after treatment with Tixel.
  each patient will be treated with the 2 modes of treatments - 2 arms in symmetrical locations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- topical treatment (Other): Topical Betamethasone for the Treatment of Vitiligo Disease
  Interventions: Other: Topical treatment
- Enhanced Transcutaneous Delivery (Experimental): Enhanced Transcutaneous Delivery of Topical Betamethasone after a treatment with Tixel device for the Treatment of Vitiligo Disease
  Interventions: Other: Enhanced Transcutaneous Delivery of Topical Betamethasone after the treatment with Tixel

INTERVENTIONS:
Other: Enhanced Transcutaneous Delivery of Topical Betamethasone after the treatment with Tixel — Tixel Parameters: exposure time 6-8 milliseconds, 400-600 μm protrusion
  Arms: Enhanced Transcutaneous Delivery
Other: Topical treatment — betamethasone ointment treatment once per day
  Arms: topical treatment

SUMMARY:
Vitiligo is the commonest acquired depigmenting disorder characterized by loss of melanocytes from the basal layer of skin causing white patches which leads to great psychological distress in many patients. Even though the pathogenic mechanisms of the loss of melanocytes are well researched, a permanent cure for the disease is still elusive. The key principle in the management of vitiligo is to attain stability and to induce active residual melanocytes to repopulate within the depigmented patch thus resulting in repigmentation. In recent years the use of various devices for enhanced transcutaneous delivery of various topical preparations has become more and more common in Dermatology. The aim of this study is to see whether using the Tixel device to enhance the penetration of topical betamethasone can improve the effectiveness of the treatment of pigment regeneration in vitiligo.

DETAILED DESCRIPTION:
Vitiligo is a psychologically devastating disorder. The fact that it typically occurs in exposed areas (the face and hands) has a major impact on self-esteem and perception of self. While lesions are usually asymptomatic, the psychosocial impact on patients can be tremendous.

Currently available medical therapies for vitiligo are unsatisfactory and there is no FDA approved drug for the treatment of vitiligo. The perfect medication for this disease would be a topically applied formulation that can rapidly restore pigmentation without systemic absorption or cutaneous side effects.

Tixel is a novel non-laser thermo-mechanical system (Tixel, Novoxel, and Israel), that is, a registered medical device in several countries worldwide. The mechanism of action is by evaporation and thermal decomposition of stratum corneum and the dehydration of epidermis.

The aim of our study is to evaluate the clinical effectiveness and safety profile of a novel approach using an energy-based device (Tixel, Novoxel, and Israel), followed by the topical application of Bethametasone for the treatment of vitiligo.

ELIGIBILITY:
Inclusion criteria:

1. Symmetric vitiligo
2. Stable vitiligo for at least six months (< 10% change in the last 6 months)
3. Diagnosis was made clinically by a dermatologist
4. Age over 18 -70 years men and women

Exclusion criteria:

1. Non Stable vitiligo
2. Contraindications for phototherapy
3. Pregnancy or lactation
4. Lack of willingness to go to phototherapy 3 times a week for at least 6 months
5. Segmental Vitiligo
6. Phototherapy or topical therapy for vitiligo in the last 1 month.

Exit criteria:

1. Intolerable to the the study treatment
2. Lack of patient's compliance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient's global impression of change (PGIC) scale | up to 2 years
  The self-report measure Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment. Although widely used in chronic pain clinical trials, PGIC's validity has not been formally assessed. PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "1- very much improved," "2- much improved," "3- minimally improved," "4-no change," "5- minimally worse," "6- much worse," or "7- very much worse."
Dermatology life quality index (DLQI) | up to 2 years
  The Dermatology life Quality Index (DLQI) is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person.
  There are 10 questions, covering the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, treatment. Each question refers to the impact of the skin disease on the patient's life over the previous week Each question is scored from 0 to 3, giving a possible score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).
  A series of validated "band descriptors" were described in 2005 to give meaning to the scores of the DLQI.
  These bands are as follows: 0-1 = No effect on patient's life, 2-5 = Small effect, 6-10 = Moderate effect, 11-20 = Very large effect, 21-30 = Extremely large effect.
Physician's global assessment (PGA) scale | up to 2 years
  0-4 scale of improvement 0- Absent: 0%
  1. Minimal: < 25%
  2. Mild: 26-50%
  3. Moderate: 51-75% 4 -Marked to complete: > 75%.

CONTACTS AND LOCATIONS:
Overall Officials: Mor Pavlovski, MD, Principal Investigator — Sourasky Medical Center
Locations (1):
- Department of Dermatology, Tel Aviv Sourasky medical center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No